CLINICAL TRIAL: NCT00002078
Title: Phase I Study of Alferon N Injection in Persons With Asymptomatic Human Immunodeficiency Virus (HIV) Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Purdue Frederick (Industry)
Collaborators: Walter Reed Army Institute of Research (WRAIR) (U.S. Federal Agency); Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Purpose: Treatment
Other Study IDs: 082A
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1993-11

CONDITIONS: HIV Infections
Keywords: Drug Evaluation; Interferon-alpha
MeSH Terms: conditions — HIV Infections | interventions — Interferon Alfa-n3

INTERVENTIONS:
Drug: Interferon alfa-n3

SUMMARY:
To determine the safety and tolerance of subcutaneous injections of natural interferon alpha (IFN) in asymptomatic HIV-positive persons and record its effects on the HIV virus in these individuals.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV-1 seropositivity.
* CD4 count > 400/mm3.
* Eligibility for care in the military medical system.

Prior Medication:

Allowed:

* Acyclovir.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* AIDS- or ARC-defining condition (unexplained weight loss, fever, diarrhea, night sweats).
* Evidence of AIDS dementia.
* Chronic hepatitis with severe liver dysfunction.
* Active gastrointestinal, renal, respiratory, endocrine, hematologic, cardiovascular, or psychiatric disorder that would limit ability to complete the study.
* Hemophilia.
* Co-existent disease likely to result in death within the next 2 years.
* Known hypersensitivity to human interferon alpha.
* Known anaphylactic hypersensitivity to mouse immunoglobulin (IgG), egg protein, or neomycin.

Concurrent Medication:

Excluded:

* Any other concurrent experimental medications.

Patients with the following prior conditions are excluded:

* History of AIDS- or ARC-defining condition (unexplained weight loss, fever, diarrhea, night sweats).
* Evidence of chronic hepatitis with severe liver dysfunction.

Prior Medication:

Excluded within 5 days prior to study entry:

* Immunosuppressive agents.
* Chemotherapy.
* Steroids.

Excluded within 45 days prior to study entry:

* BCG vaccine.
* Isoprinosine.
* Other immune modulators.

Excluded within 3 months prior to study entry:

* Any form of interferon.
* Antiviral therapy.
* Immunoregulatory therapy (other than acyclovir).

  1. Active drug abuse (narcotic or alcohol abuse documented within the past 6 months).
* Unlikely or unable to comply with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Walter Reed Army Institute of Research, Washington D.C., District of Columbia
  - Natl Naval Med Ctr, Bethesda, Maryland

REFERENCES:
- [Background] Skillman DR, Wagner K, Malone JL, Decker C, Paparello S, Meltzer MS. Phase 1 study of interferon alfa-N3 in asymptomatic HIV-infected persons. Int Conf AIDS. 1993 Jun 6-11;9(1):468 (abstract no PO-B26-1998)